CLINICAL TRIAL: NCT03423641
Title: Safety of Direct-Acting Antiviral Medications for Hepatitis C
Brief Title: An Observational Study of the Safety of Direct-acting Antivirals in Patients With Hepatitis C
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: OneFlorida Clinical Research Consortium (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Elizabeth A. McGlynn, Vice President, Kaiser Permanente Research; Executive Director, Center for Effectiveness and Safety Research, Kaiser Permanente
Other Study IDs: RI-RCR-1000
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Results first posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Hepatitis C, Chronic
Keywords: Drug-Related Side Effects and Adverse Reactions; Antiviral Agents / Adverse Effects; Antiviral Agents / Toxicity; Simeprevir; Sofosbuvir; Ledipasvir; Ombitasvir; Paritaprevir; Ritonavir; Dasabuvir; Daclatasvir; Elbasvir; Grazoprevir; Velpatasvir; Ribavirin
MeSH Terms: conditions — Hepatitis C, Chronic; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (2):
- Direct Acting Antivirals: Patients who receive a direct acting antiviral enter the DAA cohort at the time of initiation of the drug.
  Interventions: Drug: Direct Acting Antivirals
- Comparison: The exposure time of patients who have not received a direct acting antiviral (patients can change from the comparison to the DAA group once they receive the medication)

INTERVENTIONS:
Drug: Direct Acting Antivirals — The time period during which a patient is dispensed the medication and for up to 180 days after initiation of the medication.
  Groups: Direct Acting Antivirals

SUMMARY:
The investigators will assess whether patients with the Hepatitis C virus (HCV) who are prescribed direct-acting antiviral (DAA) medications experience higher rates of adverse events than patients with HCV who are untreated. The investigators hypothesize that patients receiving DAAs do not experience higher rates of adverse events compared to patients who have not received DAAs. The study population is adults between the ages of 18 and 88 with any indication of a diagnosis of HCV. An intervention group (those receiving a DAA) and comparison group (those who are not treated) will be created using medication dispensing data. Eligibility for the study will be determined from January 1, 2011 through December 31, 2017. Covariates will be collected from January 1, 2011 through December 31, 2017. Individual study sites may have access to historical data prior to 2011 that can be used as covariates or to identify individuals with HCV. The primary outcomes of interest include acute myocardial infarction, neurological outcomes (e.g. acute stroke, intracranial bleed), acute kidney failure, acute on chronic liver failure, hepatic decompensation, multiple organ dysfunction syndrome, cancer, bradyarrhythmia, and death. The secondary outcomes include decompensated cirrhosis, hospitalization, emergency department visit, and arrhythmia. Outcomes will be assessed from January 1, 2011 through December 31, 2017. The investigators will use two different analytic approaches to answer the question of interest: a Poisson regression model and marginal structural modeling (MSM). The simpler Poisson model is an extension of tabular rate of event analysis. The more complicated MSM model incorporates modeling of the treatment decision to more flexibly control for confounding by indication. For each outcome, the investigators will only record the first date an outcome occurs. Each outcome will be modeled separately.

ELIGIBILITY:
Inclusion Criteria:

* HCV viral load
* HCV genotype
* HCV qualitative
* HCV antibody
* HCV drug
* Continuously enrolled 12 months

Exclusion Criteria:

* Each outcome will be analyzed separately as time to first event, thus people who experience an outcome prior to their study start date are ineligible for analyses related to that particular outcome.

The results will be examined for sensitivity to the following possible exclusion criteria:

* Achieved SVR-12 prior to index date
* HCV treatment experienced prior to index date
* No visit in GI, Infectious Disease, or Liver Transplant / Hepatology
* No positive HCV test (genotype, viral load, or qualitative)
* No recent positive HCV test (genotype, viral load or qualitative)

Ages: 18 Years to 88 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The groups/cohorts will consist of all HCV patients from Kaiser Permanente Southern California region, Kaiser Permanente Northern California region, and the OneFlorida Clinical Research Consortium.
Sampling Method: Probability Sample
Enrollment: 33808 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A McGlynn, PhD, Principal Investigator — Kaiser Permanente

IPD SHARING:
Plan to Share IPD: Undecided
Current plan is to make a de-identified data set available to investigators under specified conditions.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a retrospective observational study, thus patients are not assigned and no one is excluded from the study after they become eligible.
Period: Overall Study
Arm/Group | Direct Acting Antivirals | Comparison
Started | 15524 | 18284
Completed | 15193 | 10210
Not Completed | 331 | 8074

BASELINE CHARACTERISTICS:
Population: There is no difference between the number of baseline participants and the numbers in participant flow.
Groups:
- Total: Total of all reporting groups
Arm/Group | Direct Acting Antivirals | Comparison | Total
Number analyzed (Participants) | 15524 | 18284 | 33808
Age, Categorical [Count of Participants; unit: Participants] — Population: There is no difference between the baseline population and the analysis population.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 12349 | 14638 | 26987
    >=65 years | 3175 | 3646 | 6821
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6092 | 6962 | 13054
  Male | 9432 | 11322 | 20754
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 112 | 116 | 228
  Asian | 891 | 772 | 1663
  Native Hawaiian or Other Pacific Islander | 49 | 51 | 100
  Black or African American | 2699 | 3838 | 6537
  White | 8670 | 9892 | 18562
  More than one race | 700 | 720 | 1420
  Unknown or Not Reported | 2403 | 2895 | 5298
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15524 | 18284 | 33808

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Acute Myocardial Infarction (AMI)
Description: Inpatient encounter with an ICD-9 diagnosis code of 410.xx or ICD-10 diagnosis code of I21.xx.
Time Frame: Patient diagnoses collected from encounters will be examined through study completion, or up to 180 days from the day the patient initiated a DAA.
Population: The analysis population consists of the subset of patients without a prior diagnosis of MI.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person years
Arm/Group | Direct Acting Antivirals | Comparison
Number analyzed (Participants) | 14959 | 17421
Events per 1000 person years | 3.3 [2.0 to 4.7] | 5.2 [4.6 to 5.8]
Statistical Analysis 1: Comparison: Direct Acting Antivirals vs Comparison; Test type: Superiority; p = .68, Marginal Structural Model; Odds Ratio (OR) = .81, 95% CI 2-sided [0.30 to 2.20] — The numerator represents the DAA group while the denominator represents the comparison group for the odds ratio

2. Primary Outcome: Incidence of Acute on Chronic Liver Failure
Description: An acute change in MELD (model for end stage liver disease) score of 5 or more and the change is deemed to have persisted (defined as meeting one of the following criteria: MELD continues to be elevated 3 months later, liver transplant, death). The minimum value for the MELD is 6.43, but there is no maximum value. Higher scores mean a worse outcome.
Time Frame: Labs and diagnoses collected from clinical encounters will be examined through study completion, or up to 180 days from the day the patient initiated a DAA.
Population: The analysis population consists of the subset of patients with MELD scores less than 15 at baseline.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person years
Arm/Group | Direct Acting Antivirals | Comparison
Number analyzed (Participants) | 13321 | 13716
Events per 1000 person years | 16.5 [13.3 to 19.7] | 24.1 [22.8 to 25.5]
Statistical Analysis 1: Comparison: Direct Acting Antivirals vs Comparison; Test type: Superiority; p = 0.01, Marginal Structural Model; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.56 to 0.91] — The numerator represents the DAA group while the denominator represents the comparison group for the odds ratio

3. Primary Outcome: Incidence of Acute Kidney Failure (AKF)
Description: Encounters with an ICD-9 diagnosis code of 584.xx or ICD-10 diagnosis code of N17.xx.
Time Frame: as for outcome 1
Population: The analysis population consists of the subset of patients without a prior diagnosis of AKF.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person years
Arm/Group | Direct Acting Antivirals | Comparison
Number analyzed (Participants) | 14321 | 16926
Events per 1000 person years | 24.2 [20.5 to 28.0] | 33.7 [32.2 to 35.2]
Statistical Analysis 1: Comparison: Direct Acting Antivirals vs Comparison; Test type: Superiority; p = 0.39, Marginal Structural Model; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.75 to 1.12] — The numerator represents the DAA group while the denominator represents the comparison group for the odds ratio

4. Primary Outcome: Incidence of Multiple Organ Dysfunction Syndrome (MODS)
Description: Inpatient encounters with ICD-9 diagnosis code of 995.92, 995.94, 785.52 or ICD-10 code of R65.11 or R65.2x.
Time Frame: as for outcome 1
Population: The analysis population consists of the subset of patients without a prior diagnosis of MODS.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person years
Arm/Group | Direct Acting Antivirals | Comparison
Number analyzed (Participants) | 15107 | 17763
Events per 1000 person years | 9.7 [7.4 to 12.0] | 17.2 [16.2 to 18.3]
Statistical Analysis 1: Comparison: Direct Acting Antivirals vs Comparison; Test type: Superiority; p = 0.01, Marginal Structural Model; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.49 to 0.90] — The numerator represents the DAA group while the denominator represents the comparison group for the odds ratio

5. Primary Outcome: Death
Description: Date of death in one or more records. Death data comes from medical records, Social Security, or state databases.
Time Frame: Death dates will be examined through study completion, or up to 180 days from the day the patient initiated a DAA.
Population: The analysis population is equivalent to the baseline population.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person years
Arm/Group | Direct Acting Antivirals | Comparison
Number analyzed (Participants) | 15524 | 18284
Events per 1000 person years | 10.7 [8.3 to 13.1] | 33.7 [32.3 to 35.1]
Statistical Analysis 1: Comparison: Direct Acting Antivirals vs Comparison; Test type: Superiority; p < 0.01, Marginal Structural Model; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.30 to 0.59] — The numerator represents the DAA group while the denominator represents the comparison group for the odds ratio

6. Primary Outcome: Incidence of Ischemic Stroke
Description: Inpatient encounters with ICD-9 diagnosis code of 433.xx, 434.xx or ICD-10 code of I63.xx, I65.xx.
Time Frame: as for outcome 1
Population: The analysis population consists of the subset of patients without a prior diagnosis of a stroke.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person years
Arm/Group | Direct Acting Antivirals | Comparison
Number analyzed (Participants) | 14758 | 17142
Events per 1000 person years | 3.6 [2.2 to 5.1] | 5.8 [5.1 to 6.4]
Statistical Analysis 1: Comparison: Direct Acting Antivirals vs Comparison; Test type: Superiority; p = 0.12, Marginal Structural Model; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.42 to 1.10] — The numerator represents the DAA group while the denominator represents the comparison group for the odds ratio

7. Primary Outcome: Incidence of Hemorrhagic Stroke
Description: Inpatient encounters with ICD-9 diagnosis code of 430.xx-432.xx or ICD-10 code of I60.xx-I62.xx
Time Frame: as for outcome 1
Population: The analysis population consists of the subset of patients without a prior diagnosis of a stroke.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person years
Arm/Group | Direct Acting Antivirals | Comparison
Number analyzed (Participants) | 14802 | 17098
Events per 1000 person years | 1.5 [0.6 to 2.3] | 3.1 [2.6 to 3.5]
Statistical Analysis 1: Comparison: Direct Acting Antivirals vs Comparison; Test type: Superiority; p = 0.34, Marginal Structural Model; Odds Ratio (OR) = 0.61, 95% CI 2-sided [0.22 to 1.70] — The numerator represents the DAA group while the denominator represents the comparison group for the odds ratio

8. Primary Outcome: Incidence of Decompensated Cirrhosis
Description: A patient will be characterized as having decompensated cirrhosis from an encounter indicating jaundice (ICD-9 diagnosis code of 782.4 or ICD-10 code of R17), ascites (ICD-9 diagnosis code of 789.5, 789.51, 789.59 or ICD-10 diagnosis code of R18.0, R18.8, K71.51, K70.11, or K70.31), or varices (ICD-9 diagnosis code of 456.0, 456.20 or ICD-10 diagnosis code of I85.01 or I85.11, or a medication dispense of lactulose or rifaximin along with a diagnosis of cirrhosis.
Time Frame: as for outcome 1
Population: The analysis population consists of the subset of patients without prior diagnosis of jaundice, ascites, hemorrhagic varices or medication dispense of lactulose or rifaximin.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person years
Arm/Group | Direct Acting Antivirals | Comparison
Number analyzed (Participants) | 13496 | 16465
Events per 1000 person years | 23.8 [20.0 to 27.7] | 38.6 [37.0 to 40.2]
Statistical Analysis 1: Comparison: Direct Acting Antivirals vs Comparison; Test type: Superiority; p < 0.01, Marginal Structural Model; Marginal Structural Model = 0.61, 95% CI 2-sided [0.49 to 0.76] — The numerator represents the DAA group while the denominator represents the comparison group for the odds ratio

9. Primary Outcome: Rate of Hospitalizations
Description: An encounter in which the place of service is an inpatient hospitalization.
Time Frame: Hospitalizations will be examined through study completion, or up to 180 days from the day the patient initiated a DAA.
Population: The analysis population is the same as the baseline population.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person years
Arm/Group | Direct Acting Antivirals | Comparison
Number analyzed (Participants) | 15524 | 18284
Events per 1000 person years | 162.8 [157.9 to 167.7] | 325.0 [320.6 to 329.4]
Statistical Analysis 1: Comparison: Direct Acting Antivirals vs Comparison; Test type: Superiority; p < 0.01, Poisson Regression; Rate Ratio = 0.71, 95% CI 2-sided [0.60 to 0.84] — The numerator represents the DAA group while the denominator represents the comparison group for the rate ratio

10. Primary Outcome: Rate of Emergency Department Visits
Description: An encounter in which the place of service is an emergency department or urgent care center.
Time Frame: ED visits will be examined through study completion, or up to 180 days from the day the patient initiated a DAA.
Population: The analysis population is the same as the baseline population.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person years
Arm/Group | Direct Acting Antivirals | Comparison
Number analyzed (Participants) | 15524 | 18284
Events per 1000 person years | 551.2 [542.3 to 560.2] | 853.4 [846.2 to 860.5]
Statistical Analysis 1: Comparison: Direct Acting Antivirals vs Comparison; Test type: Superiority; p < 0.01, Poisson Regression; Rate Ratio = 0.82, 95% CI 2-sided [0.77 to 0.87] — The numerator represents the DAA group while the denominator represents the comparison group for the rate ratio

11. Primary Outcome: Incidence of Arrhythmia
Description: Inpatient encounters with an ICD-9 diagnosis code of 427.1, 427.42, 427.5, 427.9 or an ICD-10 diagnosis code of I47.2, I49.01, I49.02, I46.9, I49.9.
Time Frame: as for outcome 1
Population: The analysis population consists of the subset of patients without a past diagnosis of arrhythmia.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person years
Arm/Group | Direct Acting Antivirals | Comparison
Number analyzed (Participants) | 13396 | 15272
Events per 1000 person years | 3.2 [1.8 to 4.5] | 4.7 [4.1 to 5.2]
Statistical Analysis 1: Comparison: Direct Acting Antivirals vs Comparison; Test type: Superiority; p = 0.02, Marginal Structural Model; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.25 to 0.88] — The numerator represents the DAA group while the denominator represents the comparison group for the odds ratio

12. Primary Outcome: Incidence of Liver Cancer
Description: Encounters with ICD-9 diagnosis code of 155.xx or ICD-10 code of C22.xx.
Time Frame: as for outcome 1
Population: The analysis population consists of the subset of patients without a prior diagnosis of liver cancer.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person years
Arm/Group | Direct Acting Antivirals | Comparison
Number analyzed (Participants) | 14905 | 17989
Events per 1000 person years | 9.3 [7.0 to 11.5] | 14.9 [13.9 to 15.8]
Statistical Analysis 1: Comparison: Direct Acting Antivirals vs Comparison; Test type: Superiority; p = 0.07, Marginal Structural Model; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.37 to 1.03] — The numerator represents the DAA group while the denominator represents the comparison group for the odds ratio

13. Primary Outcome: Incidence of Cancers Other Than Liver Cancer
Description: Encounters with ICD-9 codes 140.xx through 208.xx, except 155.xx or ICD-10 coes C00-C97 except C22.xx.
Time Frame: as for outcome 1
Population: The analysis population consists of the subset of patients without a prior diagnosis of cancer.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person years
Arm/Group | Direct Acting Antivirals | Comparison
Number analyzed (Participants) | 13254 | 16689
Events per 1000 person years | 20.7 [17.1 to 24.3] | 26.4 [25.0 to 27.7]
Statistical Analysis 1: Comparison: Direct Acting Antivirals vs Comparison; Test type: Superiority; p = 0.11, Marginal Structural Model; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.63 to 1.05] — The numerator represents the DAA group while the denominator represents the comparison group for the odds ratio

14. Primary Outcome: Incidence of HBV Reactivation
Description: We identified HBV reactivations in three different ways [Di Bisceglie et al., 2015; Yanny et al., 2018]: (1) patients who had a history of Hepatitis B core antibody (HBcAb) positive and were Hepatitis B surface antigen (HBsAg) negative at the time of initiating DAA therapy who became HBsAg positive within 180 days after receiving a DAA; (2) patients with undetectable levels of HBV DNA at the time of initiating DAA therapy who had a numerical result within 180 days after receiving a DAA; (3) patients with a numerical HBV DNA result at the time of initiating DAA therapy whose viral load increased by a factor of 10 within 180 days after receiving a DAA. For all methods of detecting a reactivation, we required that the reactivations be clinically significant: bilirubin at least 3, aspartate aminotransferase (AST) at least 400, or alanine aminotransferase (ALT) at least 500.
Time Frame: Labs will be for up to 180 days following the initiation of a DAA.
Population: At the time of initiating DAA therapy, at least one of the following had to be true (1) Hepatitis B core antibody (HBcAb) positive and Hepatitis B surface antigen (HBsAg) negative (2) Hepatitis B core antibody (HBcAb) positive and undetectable levels of HBV DNA; (3) numerical HBV DNA result
Measure: Count of Participants; unit: Participants
Arm/Group | Direct Acting Antivirals
Number analyzed (Participants) | 2308
Participants | 1

ADVERSE EVENTS:
Time Frame: This was a retrospective observational study, so any adverse event data would have been collected during contact with a medical provider.
Description: This was a retrospective observational study. Any adverse event reporting would have been the responsibility of the medical provider. We did not seek out adverse event information above and beyond the outcomes of interest in our study.
Arm/Group | Direct Acting Antivirals | Comparison
All-Cause Mortality (participants affected / at risk) | 77/15524 | 2186/18284
Serious Adverse Events (participants affected / at risk) | 0/15524 | 0/18284
Other Adverse Events (participants affected / at risk) | 0/15524 | 0/18284

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/41/NCT03423641/SAP_000.pdf
  • Study Protocol (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT03423641/Prot_001.pdf